CLINICAL TRIAL: NCT01598363
Title: An Open-Label Study of the Effect of Bardoxolone Methyl on the Single Dose Pharmacokinetics of Digoxin and Rosuvastatin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 402-C-1104
Record Dates: First submitted 2012-05-11; First posted 2012-05-15 (Estimated); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Digoxin; Rosuvastatin Calcium

ARMS (2):
- Digoxin 0.5mg, Bardoxolone Methyl 20mg and 60mg (Experimental)
  Interventions: Drug: Digoxin
- Rosuvastatin 20mg, Bardoxolone Methyl 20mg and 60mg (Experimental)
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Digoxin — Oral, Day 1 and Day 10
  Arms: Digoxin 0.5mg, Bardoxolone Methyl 20mg and 60mg
Drug: Rosuvastatin — Oral, Day 1 and Day 10
  Arms: Rosuvastatin 20mg, Bardoxolone Methyl 20mg and 60mg

SUMMARY:
The purpose of this study is to evaluate the potential effect of bardoxolone methyl on the pharmacokinetics of digoxin and rosuvastatin and to assess the safety of the concomitant administration of bardoxolone methyl with digoxin or rosuvastatin.

DETAILED DESCRIPTION:
Subjects in Cohort 1 will receive a single dose of digoxin (0.5 mg) on Study Day 1, an initial dose of bardoxolone methyl (60 mg) and a single dose of digoxin (0.5 mg) on Study Day 10, and once daily doses of bardoxolone methyl (20 mg) on Study Days 11 through 14. Subjects in Cohort 2 will receive a single dose of rosuvastatin (20 mg) on Study Day 1, an initial dose of bardoxolone methyl (60 mg) and a single dose of rosuvastatin (20 mg) on Study Day 10, and once daily doses of bardoxolone methyl (20 mg) on Study Days 11 through 14. All doses will be given in the morning under fasting conditions. Bardoxolone methyl and the probe substrates (digoxin, rosuvastatin) will be dosed at the same time. Confinement will begin on Study Day -1 (Study Day before the first dosing day) and end after the collection of the 216 hour blood samples and scheduled study procedures on Study Day 19.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between 18 and 45 years, inclusive;
* Willing to practice a method of birth control (both males who have partners of childbearing potential and females of childbearing potential) during screening, while taking study drug, and for at least 30 days after the last dose of study drug is ingested;
* Body mass index (BMI) between 19 and 31 kg/m2, inclusive;
* Willing and able to give written informed consent for study participation;
* Willing and able to cooperate with all aspects of the protocol.

Exclusion Criteria:

* Participated in another clinical trial of an investigational drug (or medical device) within 30 days before Study Day -1, or are currently participating in another trial of an investigational drug (or medical device);
* Any condition possibly affecting absorption, distribution, metabolism or excretion of drugs that may confound the analyses conducted in this study (for example: previous surgery on the gastrointestinal tract that includes removal of parts of stomach, bowel, liver, gall bladder, pancreas, venacaval shunts, or transjugular intrahepatic portosystemic shunts);
* Known hypersensitivity to any component in the formulation of bardoxolone methyl, LANOXIN®, or CRESTOR®;
* Evidence or history of or concurrent clinically significant allergic (except for untreated, asymptomatic, seasonal allergies at time of dose administration), hematological, endocrine, immunological, renal, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease that in the judgment of the investigator could potentially either pose a health risk to the subject during the study or influence the study outcome;
* Evidence of hepatic or biliary dysfunction including elevation of total bilirubin, direct bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma glutamyl transpeptidase (GGT), lactate dehydrogenase (LDH), or alkaline phosphatase levels to greater than the upper limit of normal (ULN);
* Positive test results for human immunodeficiency virus type 1 or 2 antibody, hepatitis B surface antigen, or hepatitis C virus antibody at screening;
* Any medical or dental procedure, no matter how minor, that is planned or anticipated to occur during the conduct of the study;
* History of alcohol abuse or dependence within the last year;
* Any vaccination within 30 days before start of this study and throughout the study;
* Use of aspirin, non-steroidal anti-inflammatory agents, or acetaminophen within 5 days before Study Day 1; use of aspirin or non-steroidal anti-inflammatory agents (but not acetaminophen) will be allowed for isolated episodes of pain at the discretion of the investigator;
* Use of or need for any systemic drug(s) including vitamins or herbal preparations other than drugs used for contraception, within 30 days before entry into the study or during the study;
* Donation or receipt of blood or blood components within the 4 weeks before Study Day -1, The investigator should instruct subjects who participate in this study not to donate blood or blood components for 4 weeks after the completion of the study;
* Any diagnostic or intervention procedure requiring a contrast agent within the 30 days before study participation;
* Systolic blood pressure > 140mmHg or < 100mmHg or a diastolic blood pressure >95 mmHg at screening measured after 5 minutes in a sitting position;
* A pulse rate at rest in a sitting position of < 50 bpm or > 100 bpm;
* Abnormal screening ECG (including a QTcF interval of >450 ms) which is interpreted by the investigator to be clinically significant, or any clinical evidence of Wolff-Parkinson-White syndrome, intermittent complete heart block, second degree heart block or prolonged PR interval of ≥ 200 msec on the 12-lead ECG;
* Use of tobacco- or nicotine-containing products (that is, cigarettes, cigars, chewing tobacco, snuff, etc) or products for smoking cessation within 2 weeks before Study Day -1;
* Consumed alcohol or xanthine-containing products (e.g., tea, coffee, chocolate, cola, etc.) within 72 hours before Study Day -1;
* Treated with any investigational agent within 30 days before Study Day -1, 5 half-lives or twice the duration of biological effect of the previous investigational drug (whichever is longer);
* A history of drug abuse or who test positive for drug(s) of abuse (ethanol, amphetamines, benzodiazepines, barbiturates, cocaine, opiates, or cannabinoids) or cotinine (indicating active current smoking) at the screening or Study Day -1;
* Female subjects who are planning a pregnancy or are pregnant or lactating;
* Deemed by the investigator to be inappropriate for this study, including subjects who are unable to communicate with the investigator due to language problems, poor mental development, or impaired cerebral function.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-06-30 (Actual); Primary Completion 2012-07-31 (Actual); Study Completion 2012-07-31 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  For Digoxin and Rosuvastatin

SECONDARY OUTCOMES:
Time to maximum observed concentration | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  For Digoxin and Rosuvastatin
Area under the plasma-concentration time-curve | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  For Digoxin and Rosuvastatin
Oral clearance | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  For Digoxin and Rosuvastatin
Terminal rate constant | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  For Digoxin and Rosuvastatin
Terminal half-life | 0, 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216 hours post-dose
  For Digoxin and Rosuvastatin
Amount excreted in Urine | 0-24, 24-48, 484-72, 72-96, 96-120, 120-144, 144-168, 168-192, 192-216 hours post-dose
  For Digoxin only
Fraction of the dose excreted in Urine | 0-24, 24-48, 484-72, 72-96, 96-120, 120-144, 144-168, 168-192, 192-216 hours post-dose
  For Digoxin only
Renal clearance | 0-24, 24-48, 484-72, 72-96, 96-120, 120-144, 144-168, 168-192, 192-216 hours post-dose
  For Digoxin only
Number of patients with Adverse Events | Approximately 1 year
Determination of concentration for Bardoxolone Methyl | 0 hours and 3 hours after dosing
  Sample will be taken at 0 hours and 3 hours after dosing only on Study Days 10, 12 and 14

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Clinical Research, LLC, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/